CLINICAL TRIAL: NCT01868529
Title: A Randomised, Single Centre, Double-blind, Two-Period Cross-over, Multiple Dose Trial Comparing the Pharmacodynamic Response of Insulin 454 With Insulin Glargine at Steady-State Conditions in Subjects With Type 1 Diabetes Mellitus
Brief Title: Comparison of Insulin Degludec With Insulin Glargine in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1876; 2007-003534-41 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine
- Medium dose (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine
- High dose (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Once daily dosing administered subcutaneously (s.c., under the skin) followed by a clamp visit. The two treatment periods will be separated by a wash-out period where the subjects will resume their normal insulin treatment.
Drug: insulin glargine — Once daily dosing administered subcutaneously (s.c., under the skin) followed by a clamp visit. The two treatment periods will be separated by a wash-out period where the subjects will resume their normal insulin treatment.

SUMMARY:
This trial was conducted in Europe. The aim of this trial was to compare the pharmacodynamic (the effect of the investigated drug on the body) response of insulin degludec (insulin 454) with insulin glargine at steady-state conditions in subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) and treated with insulin for at least 12 months
* Subject is considered to be generally healthy, except for the underlying diabetes mellitus and related morbidity (such as well controlled hypertension and dyslipidaemia) based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
* Body Mass Index (BMI) between 18.0 and 28.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin (HbA1c) below or equal to 10.0 % based on central laboratory results
* Subject with a daily basal insulin requirement of between 0.2 IU/kg/day and 0.6 IU/kg/day will be allowed to participate in the trial. Current total daily treatment with insulin must be less than 1.2 U/kg/day

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Subject who has participated in any other trials involving investigational products within 3 months preceding the start of dosing
* Subject who has donated any blood or plasma in the past month or in excess of 500 mL within the 12 weeks preceding screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | 0-24 hours in steady-state

SECONDARY OUTCOMES:
Area under the serum insulin concentration curve at steady state | 0-24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com